CLINICAL TRIAL: NCT03537417
Title: Changes in Heart Rate Variability in Ventilated Patients Undergoing Tension Pneumothorax for Thoracoscopic Cervical Sympathectomy
Brief Title: Heart Rate Variability in Pneumothorax
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Dr. Amit Lehavi MD FANZCA, Director of Pediatric Anesthesia, Rambam Health Care Campus
Other Study IDs: RMB 144-18
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tension pneumothorax group: Patients undergoing intentional pneumothorax for thoracoscopic ablation of cervical sympathetic chain as a treatment for hyperhidrosis
  Interventions: Procedure: for thoracoscopic ablation of cervical sympathetic chain

INTERVENTIONS:
Procedure: for thoracoscopic ablation of cervical sympathetic chain — bilateral thoracoscopic ablation of cervical sympathetic chain as a treatment for hyperhidrosis

SUMMARY:
Changes in heart rate variability in anesthetized, ventilated patients undergoing tension pneumothorax for thoracoscopic cervical sympathectomy

ELIGIBILITY:
Inclusion Criteria:

* age 15 - 50 years
* body mass index 25 - 45

Exclusion Criteria:

* heart rate other than sinus
* cardiac pacemaker status
* heart transplant

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients undergoing tension pneumothorax for thoracoscopic cervical sympathectomy for hyperhidrosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in heart rate variability | From immediately after induction of general anesthesia and mechanical ventilation to 10 minutes after initiation of pneumothorax
  Non linear changes in R-R intervals extracted from ECG